CLINICAL TRIAL: NCT01638507
Title: Resolute Integrity US A Postapproval Study of the Medtronic Resolute™ Integrity Zotarolimus-Eluting Coronary Stent System in the Treatment of De Novo Lesions in Native Coronary Arteries With a Reference Vessel Diameter of 2.25 mm to 4.2 mm
Brief Title: An Evaluation of the Commercially Available Medtronic Resolute Integrity Zotarolimus-Eluting Coronary Stent System
Acronym: RI-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP 126
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Disease
Keywords: TARGET LESION REVASCULARIZATION (TLR); TARGET VESSEL REVASCULARIZATION (TVR); Coronary Artery Disease; MYOCARDIAL INFARCTION (MI); PERCUTANEOUS CORONARY INTERVENTION (PCI); STENT THROMBOSIS; TARGET LESION FAILURE (TLF)
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resolute Integrity (Other): Medtronic Resolute Integrity Zotarolimus-Eluting Coronary Stent System (Resolute Integrity Stent)
  Interventions: Device: Resolute Integrity Stent

INTERVENTIONS:
Device: Resolute Integrity Stent — Medtronic Resolute Integrity Zotarolimus-Eluting Coronary Stent System

SUMMARY:
The purpose of this post approval study is to conduct a prospective, multicenter evaluation of the procedural and clinical outcomes of subjects that are treated with the commercially available Medtronic Resolute Integrity Zotarolimus-Eluting Coronary Stent System.

DETAILED DESCRIPTION:
The purpose and objective is to assess the safety and efficacy of the Resolute Integrity Stent for the treatment of de novo lesions in native coronary arteries with a reference vessel diameter(RD) of 2.25mm to 4.2mm in two groups of patients, specifically those patients receiving stents less than or equal to 30mm in length.

ELIGIBILITY:
General and Angiographic Inclusion Criteria highlights:

* Acceptable candidate for percutaneous coronary intervention (PCI),stenting, and emergency coronary artery bypass graft surgery
* Clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia and/or positive functional study
* Informed consent
* Patient agrees to comply with specified follow-up evaluations
* Single target lesion or two target lesions located in separate coronary arteries
* De novo lesion(s) in native coronary artery(ies)
* Target lesion(s) ≤ 27 mm in length
* Target vessel(s) have reference vessel diameter 2.25 mm to 4.2 mm

General and Angiographic Exclusion Criteria highlights:

* Within 7 days of index procedure platelet count <100,000 cells/mm³ or >700,000 cells/mm³; White Blood Cell (WBC) count <3,000 cells/mm³; serum creatinine level >2.5 mg/dl
* Acute MI within 72 hrs of the intended trial procedure (QWMI or any elevation of Creatine Kinase-MB (CK-MB) > lab upper limit of normal)
* Previous PCI of target vessel(s) within 9 months prior to the procedure
* Planned PCI of any vessel within 30 days post-index procedure and/or planned PCI of target vessel(s) within 12 months post-index procedure
* History of stroke or Transient Ischemic Attack (TIA) within prior 6 months
* Participating in investigational drug/device study that has not completed primary endpoint or interferes with study endpoints
* Inability to comply with required trial antiplatelet regimen
* Previous stent in target vessel unless it has been at least 9 months since stent placed and target lesion(s) is/are at least 15 mm from previous stent
* Target vessel(s) has/have other lesions w/ > 40% diameter stenosis
* Unprotected left main coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Caputo, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Joseph's Hospital Health Center, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 230 PEG subjects were enrolled from 29 study sites in the United States. The first subject was enrolled on July 23, 2012 and the last subject was enrolled on May 31, 2013.
Groups:
- Primary Enrollment Group (PEG): Patients with one or two de novo lesions in native coronary arteries with a reference vessel diameter (RVD) of 2.25 mm to 4.2 mm, treated with stents less than or equal to 30 mm in length.
Period: Overall Study
Arm/Group | Primary Enrollment Group (PEG)
Started | 230
Completed | 224
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- Primary Enrollment Group (PEG): Patients who have one or two de novo lesions in native coronary arteries with a reference vessel diameter (RVD) of 2.25 mm to 4.2 mm, treated with stents less than or equal to 30 mm in length.
Arm/Group | Primary Enrollment Group (PEG)
Number analyzed (Participants) | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 160

OUTCOME MEASURES:

1. Primary Outcome: Composite Rate of Cardiac Death and Target Vessel Myocardial Infarction (MI)
Time Frame: 12 months
Population: The primary analysis set was the Intent-To-Treat (ITT) population, defined as all patients who signed the written informed consent and were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Primary Enrollment Group (PEG): Patients who have one or two de novo lesions in native coronary arteries with a reference vessel diameter (RVD) of 2.25 mm to 4.2 mm, treated with stents of less than or equal to 30 mm in length.
Arm/Group | Primary Enrollment Group (PEG)
Number analyzed (Participants) | 220
percentage of participants | 3.6 [1.6 to 7.0]

2. Secondary Outcome: Composite Endpoints: Major Adverse Cardiac Events (MACE), Target Lesion Failure (TLF), Target Vessel Failure (TVF), Cardiac Death and Target Vessel MI
Time Frame: 12 months
Measure: Number; unit: percentage of composite
Arm/Group | Primary Enrollment Group (PEG)
Number analyzed (Participants) | 220
percentage of composite | 15.0

3. Secondary Outcome: Clinical Endpoint: Death
Time Frame: 12 months
Measure: Number; unit: percentage of death
Arm/Group | Primary Enrollment Group (PEG)
Number analyzed (Participants) | 220
percentage of death | 1.8

4. Secondary Outcome: Dual Antiplatelet Therapy (DAPT) Compliance
Time Frame: 12 months
Measure: Number; unit: percentage of compliance
Arm/Group | Primary Enrollment Group (PEG)
Number analyzed (Participants) | 212
percentage of compliance | 89.2

5. Secondary Outcome: Clinical Endpoint: TLR
Time Frame: 12 months
Measure: Number; unit: percentage of TLR
Arm/Group | Primary Enrollment Group (PEG)
Number analyzed (Participants) | 220
percentage of TLR | 2.3

6. Secondary Outcome: Clinical Endpoint: TVR
Time Frame: 12 months
Measure: Number; unit: percentage of TVR
Arm/Group | Primary Enrollment Group (PEG)
Number analyzed (Participants) | 220
percentage of TVR | 4.5

7. Secondary Outcome: Clinical Endpoint: MI
Time Frame: 12 months
Measure: Number; unit: percentage of MIs
Arm/Group | Primary Enrollment Group (PEG)
Number analyzed (Participants) | 220
percentage of MIs | 2.7

8. Secondary Outcome: Clinical Endpoint: ST
Time Frame: 12 months
Measure: Number; unit: percentage of ST
Arm/Group | Primary Enrollment Group (PEG)
Number analyzed (Participants) | 220
percentage of ST | 0.9

9. Secondary Outcome: Clinical Endpoint: Stroke
Time Frame: 12 months
Measure: Number; unit: percentage of strokes
Arm/Group | Primary Enrollment Group (PEG)
Number analyzed (Participants) | 220
percentage of strokes | 0.5

10. Secondary Outcome: Clinical Endpoint: Bleeding Complications in General
Time Frame: 12 months
Measure: Number; unit: percentage of bleeding complications
Arm/Group | Primary Enrollment Group (PEG)
Number analyzed (Participants) | 220
percentage of bleeding complications | 11.4

ADVERSE EVENTS:
Arm/Group | Primary Enrollment Group (PEG)
Serious Adverse Events (participants affected / at risk) | 88/230
Other Adverse Events (participants affected / at risk) | 51/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Enrollment Group (PEG) (N=230)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3)
Angina Pectoris (Cardiac disorders) | 7 (8)
Angina Unstable (Cardiac disorders) | 4 (4)
Arteriospasm Coronary (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 3 (3)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 7 (7)
Coronary Artery Dissection (Cardiac disorders) | 7 (7)
In-Stent Coronary Artery Restenosis (Cardiac disorders) | 1 (1)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 5 (5)
Sick Sinus Syndrome (Cardiac disorders) | 2 (2)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Deformity Of Orbit (Eye disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (2)
Gastrointestinal Mucosal Disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Mesenteric Artery Stenosis (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Chest Pain (General disorders) | 17 (21)
Death (General disorders) | 1 (1)
Drowning (General disorders) | 1 (1)
Implant Site Haematoma (General disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 4 (6)
Oedema Peripheral (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
In-Stent Arterial Restenosis (Injury, poisoning and procedural complications) | 2 (2)
Thrombosis In Device (Injury, poisoning and procedural complications) | 1 (1)
Cardiac Enzymes Increased (Investigations) | 2 (2)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Factitious Disorder (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Therapeutic Embolisation (Surgical and medical procedures) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 1 (1)
Arterial Haemorrhage (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Artery Dissection (Vascular disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Femoral Artery Occlusion (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Intermittent Claudication (Vascular disorders) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1)
Shock Haemorrhagic (Vascular disorders) | 1 (1)
Vascular Occlusion (Vascular disorders) | 3 (3)
Vascular Pseudoaneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Enrollment Group (PEG) (N=230)
Angina Pectoris (Cardiac disorders) | 13 (15)
Chest Pain (General disorders) | 24 (26)
Cardiac Enzymes Increased (Investigations) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For any publication or presentation of the Protected Materials or any portion thereof, a manuscript of the paper, abstract or any materials will be provided by Consultant to Sponsor for its approval at least sixty (60days) for manuscripts and thirty (30) days for presentations prior to outside submission. Medtronic shall have the right to request reasonable modifications of any manuscript or other materials to be published or presented.